**Title:** Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Sepsis Associated with Acute Necrotizing Soft Tissue Infections, The NASTI HAT Trial

**Document Date:** April 28, 2021

**Document Type:** Informed Consent Form (ICF)

# PATIENT INFORMED CONSENT/HIPAA AUTHORIZATION

Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Sepsis Associated with Acute Necrotizing Soft Tissue Infections

## **INTRODUCTION:**

You are being asked to participate in a research study since you have been diagnosed with an acute necrotizing soft tissue infection and sepsis. This study will focus on the use of an investigational treatment of hydrocortisone, ascorbic acid (vitamin C), and thiamine (vitamin B1), hereafter referred to as HAT, as a possible treatment of sepsis. Hydrocortisone is a corticosteroid commonly used in the hospital, while thiamine and ascorbic acid are both vitamins. This regimen has been used to treat patients with sepsis and one study showed a decrease in the number of deaths, but no studies have yet copied these results. Additionally, no studies have specifically examined its use in the treatment of patients with acute necrotizing soft tissue infections. The purpose of this study is to determine if treatment with HAT in patients with necrotizing soft tissue infections and sepsis results in improved survival. By participating, you will still receive the standard medical and surgical care you would have otherwise received, with the possible addition of HAT. You do not have to participate in this research study. It is important that before you make a decision to participate, you read the rest of this form. You should ask as many questions as needed to understand what will happen to you if you participate in this study.

#### **PROCEDURES:**

If you choose to participate in the study, you will be randomized to receive or not receive HAT (like the flip of a coin). The HAT medications will be given through your IV (intravenous). If you do not receive HAT, you will be given an intravenous normal saline solution (a placebo) instead. Your physician will not know which one you are receiving as part of the study. However, other than receiving or not receiving the study treatment, there will be no difference in the medical or surgical care that you receive. The pharmacy team will be aware of all your medications including the study treatment. All patients in the study will receive the same quality of care as those who are not involved. Your participation will not require you to do anything outside of receiving treatment. No follow up appointments are required for participation in this study. As a participant, data from your hospital stay will be used in the study. Data pertinent to the study will be collected and stored in a secure database. You will be included in this study until hospital discharge, when study participation ends. The study plans to enroll a total of 132 participants.

## **RISKS:**

Like any treatment, there are potential risks with the administration of HAT. Based on the available studies to date, the risks appear overall low and the treatment is generally considered safe. However, risks do exist. Furthermore, not all possible risks are listed here and as with any new treatment, some risks may be unknown at this time. Some of the more severe possible adverse reactions of each medication are listed here. Hydrocortisone can cause elevated sodium levels and gastrointestinal bleeding. There are reports of oxalate nephropathy from ascorbic acid (vitamin C) use. This is a potentially devastating condition in which calcium oxalate crystals develop in the tissue of the kidney that can cause permanent kidney damage. To our knowledge, this is rare and appears more common with higher doses and/or a longer duration of treatment with vitamin C than used in this study. Thiamine can cause gastrointestinal bleeding. Finally, as with any medication and/or vitamin, other adverse reactions can occur, including but not limited to, a severe life-threatening allergic reaction (anaphylaxis). Your physician will be monitoring you during your treatment course. If any concerns arise for an adverse event related to the study, the study treatment will be discontinued and you will be treated accordingly for the adverse event.

The potential risks due to a necrotizing soft tissue infection and sepsis are expected to be no different for you whether you are enrolled in this study or not.

If you feel that you are experiencing any bad effects from your participation in this study, you should contact Dr. Resch, Dr. Grantham, Dr. Waswick, or a member of the research team immediately.

#### PREGNANCY RELATED RISK:

If you are a woman of childbearing potential, you will have a pregnancy test as part of your normal work-up before surgery. In the event you are pregnant, you will not be allowed to participate in this study.

### **NEW FINDINGS STATEMENT:**

You will be informed if any significant new findings develop during the course of the study that may affect your willingness to participate in this study.

#### **BENEFITS:**

You may or may not benefit directly by participating in this research study. You are helping to prove that there are, or are not, benefits to treatment with HAT. Thus, you would be participating in research that could help other patients in the future.

#### **ALTERNATIVE TREATMENTS:**

There is no specific alternative treatment. If you do not participate in the study, you will still receive the standard medical and surgical care.

### **PARTICIPATION:**

Your participation in this study is voluntary. Your refusal to participate in this study will involve no penalty or loss of benefits to which you would otherwise be entitled, and you are free to stop participation at any time without penalty or loss of benefits to which you would otherwise be entitled. If you withdraw your consent, you will not be allowed to participate in this research study. By signing this consent, you acknowledge that no guarantees have been made to you as to results that may be obtained.

Your participation in this study may also be discontinued at any time, and without your consent, if in your physician's or the study team's opinion this would be in your best interest.

#### COSTS:

Participants will never be charged for study-related drugs in this study, regardless of the group to which they are randomized. This means that participation in this study will not cost you more or less than the cost of normal care. No charges for care other than those you would normally receive will be incurred during the study and the cost for your normal care will be you and/or your insurance provider's responsibility.

## **PAYMENT TO SUBJECTS:**

You will not be compensated by Ascension Via Christi Hospitals Wichita, Inc., the University of Kansas Medical Center, or other participating organizations for participation in this study.

## HOW IS THE INVESTIGATOR PAID FOR HIS WORK:

The investigators are being reimbursed for their time and costs for your normal care. Dr. Thomas Resch, the Principal Investigator of this study, is also reimbursed as part of his medical director duties for participating in burn research. Beyond those duties, there is no specific reimbursement for this research.

## IN THE EVENT OF INJURY:

In the event you experience a serious side effect during this study, you should immediately contact Dr. Thomas Resch, Dr. David Grantham, or Dr. William Waswick at (316) 268-5000.

If you have a bodily injury as a result of participating in this study, care will be provided for you at the usual charge. No financial payments or other form of compensation (such as for lost wages or discomfort) will be provided by the researchers or any of the participating organizations. Claims will be submitted to your health insurance policy, your government program, or other third party, but you will be billed for the costs of that care to the extent insurance does not cover them. You do not give up any of your legal rights by signing this form.

You should acknowledge that no guarantee has been made to you as to results that may be obtained. Ascension Via Christi Hospitals Wichita, Inc. does not provide free medical treatment or payment for injuries resulting from participation in biomedical or behavioral research.

If you believe you have been injured as a result of participating in research at Ascension Via Christi, you should contact Dr. Thomas Resch, the Principal Investigator of this study. Compensation to persons who are injured as a result of participating in research at may be available, under certain conditions, as determined by state law or the Kansas Tort Claims Act.

#### CONFIDENTIALITY AND PRIVACY AUTHORIZATION:

Efforts will be made to keep your personal information confidential. Researchers cannot guarantee absolute confidentiality. If the results of this study are published or presented in public, information that identifies you will be removed.

The privacy of your health information is protected by a federal law known as the Health Insurance Portability and Accountability Act (HIPAA). By signing this form, you are giving permission ("authorization") for Ascension Via Christi Hospitals Wichita, Inc. to use and share your health information for the purposes of this research study. If you decide not to sign the form, you cannot be in the study.

To do this research, we need to collect health information that identifies you. We will collect information from activities described in the Procedures section of this form and from your medical record.

By signing this consent, you are giving Dr. Thomas Resch, Dr. David Grantham, Dr. William Waswick, and the research team permission to share information about you with persons or groups outside of Ascension Via Christi Hospitals Wichita, Inc. Your information will be shared with officials who oversee research, including members of the Institutional Review Boards of Ascension Via Christi Hospitals Wichita, Inc. and the University of Kansas School of Medicine and other committees and offices that review and monitor research studies. Study records might be reviewed by government officials who oversee research such as the U.S. Food and Drug Administration (FDA), if a regulatory review takes place. The purpose for using and sharing your information is to make sure the study is done properly.

Once your health information has been disclosed to anyone outside of this study, the information may no longer be protected under this authorization.

You will not be allowed to review the information collected for the research study until after the study is completed. When the study is over, you will have the right to access the information.

Your permission to use and share health information will not expire unless you cancel it. Any research information that is placed in your medical record will be kept indefinitely.

## **QUESTIONS:**

In the event you have any questions, suggestions, concerns, or complaints about this study you may contact Dr. Thomas Resch, Dr. David Grantham or Dr. William Waswick at (316) 268-5000.

If you have any questions about your rights as a research subject, you may call the Ascension Via Christi Hospitals Wichita, Inc. Institutional Review Board at (316) 291-4774. If you have any questions or concerns about your privacy rights, you may call the Ascension Via Christi Hospitals Wichita, Inc. Privacy Officer at (316) 858-4945.

## SUBJECT RIGHTS AND WITHDRAWAL FROM THE STUDY:

Your participation in this study is voluntary. Your decision to not participate, or to quit at any time, can be made

Page 3 of 4 (Version 1: April 28, 2021)

without penalty or loss of benefits. Your decision not to participate or quit will have no effect upon the medical care or treatment you receive now or in the future. The entire study may be discontinued for any reason without your consent by the investigators conducting the study.

You have a right to change your mind about allowing the research team to have access to your health information. If you want to cancel permission to use your health information, you should send a written request to Dr. Thomas Resch, Dr. David Grantham, or Dr. William Waswick. The mailing address is: KUSM-W; Department of Surgery, Room 3082; 929 N. Saint Francis St.; Wichita, KS 67214. If you cancel permission to use your health information, you will be withdrawn from the study. The research team will stop collecting any additional information about you. The research team may use and share information that was gathered before they received your cancellation. Additionally, if you cancel permission, the researchers may still use your information if you have an adverse event (a bad effect).

## **CONSENT:**

A member of the research team has given you information about this research study. They have explained what will be done and how long it will take. They explained any inconvenience, discomfort, or risks that may be experienced during this study.

By signing this consent/authorization form, you indicate that you freely and voluntarily consent to participate in this research study. Further, by your signature, you indicate that you have read the information in this form and have had an opportunity to ask questions and have them answered. You will be given a signed copy of the consent form to keep for your records. If you choose not to sign this consent form, you cannot participate in this study.

| Print Subject's Name | | |
|----------------------------------------------------|---------------|------|
| Thit Subjects Name | | |
| Signature of Subject | Date | Time |
| Print Legally Authorized Representative's Name | | |
| Relationship of Authorized Representative to the S | Study Subject | |
| Signature of Legally Authorized Representative | Date | Time |
| Print Name of Person Obtaining Consent | | |
| Signature of Person Obtaining Consent | <br>Date | Time |